CLINICAL TRIAL: NCT07293559
Title: Understanding Practices of Lactation and Infant Feeding Together With Women With HIV in the United States
Acronym: UPLIFT
Status: Not yet recruiting | Type: Observational
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: University of Colorado, Denver (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: IMPAACT 2046
Record Dates: First submitted 2025-12-16; First posted 2025-12-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: HIV-1-infection; Breastfeeding; Pregnancy Related
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Core Activity 2 participants will be asked whether they agree to storage and future research testing of breastmilk specimens. Human genetic testing of leftover specimens is optional and may be declined.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Core Activity 1: This core activity aims to explore current site-level infant feeding practices and infant feeding decision-making and preferences at selected sites in the US.
  Interventions: Other: No intervention provided in this study
- Core Activity 2: This core activity aims to examine infant feeding practices and outcomes among women with HIV at selected sites in the US and to describe the financial implications of different infant feeding choices.
  Interventions: Other: No intervention provided in this study
- Core Activity 3: This core activity aims to pilot and assess the feasibility and acceptability of a national registry of breastfeeding women with HIV in the US.
  Interventions: Other: No intervention provided in this study

INTERVENTIONS:
Other: No intervention provided in this study — None; No intervention provided in this study

SUMMARY:
IMPAACT 2046/UPLIFT (Understanding Practices of Lactation and Infant Feeding decisions Together with women with HIV) is a multi-site, mixed-methods, observational cohort study. The purpose of the study is to explore infant feeding preferences, practices, and outcomes among mothers with HIV and their families in the United States. It will employ both qualitative and quantitative research methods to address existing knowledge gaps and to understand the clinical, behavioral, and social factors influencing infant feeding decisions. As part of the study's mixed method approach, a longitudinal cohort study of mothers and their infants will be established. The study also aims to pilot a national registry of breastfeeding women living with HIV in the United States.

DETAILED DESCRIPTION:
This is a convergent mixed-method, multisite study to identify factors in infant feeding decisions and explore infant feeding perspectives, preferences, practices and outcomes among women with HIV in the US. Feasibility and acceptability of developing a national registry of breastfeeding women with HIV in the US will also be assessed. The study sites will enroll women with HIV who are pregnant or postpartum (PPWH), healthcare providers (HCPs) and ancillary healthcare professionals (AHPs), other influential individuals who contribute to infant feeding decisions, and pilot registry testers.

The study will be comprised of three core activities:

* Core Activity 1: Will explore the multifaceted process of infant feeding decision-making, and describe clinical practice, and counseling approaches via in-depth interviews (IDIs) and surveys. IDIs will be completed with PPWH, influential people who contribute to infant feeding decisions, HCPs, and AHPs. HCPs and AHPs will also complete self-administered surveys, and site staff at each site will complete site-level surveys to inform a landscape analysis.
* Core Activity 2: Will establish an observational prospective cohort of PPWH, and their liveborn infants, to examine current infant feeding practices and outcomes and their associated costs and cost benefits.
* Core Activity 3: Will develop and pilot a national registry of breastfeeding women with HIV and assess its feasibility and acceptability among pilot registry testers.

ELIGIBILITY:
Core Activity 1 Inclusion Criteria: Pregnant and Postpartum Women with HIV

* Is of legal age or circumstance to provide independent informed consent
* Belongs to one of the following five categories:

  * Is pregnant with a gestational age of 28 0/7 to 37 6/7 weeks at entry and is considering breastfeeding
  * Is pregnant with a gestational age of 28 0/7 to 37 6/7 weeks at entry and is not considering breastfeeding
  * Gave birth to a live born infant after 28 February 2023, is over 4 weeks postpartum, did not breastfeed for any duration and has no intent to breastfeed
  * Gave birth to a live born infant after 28 February 2023, is over 4 weeks postpartum, breastfed for less than four weeks, and has weaned
  * Gave birth to a live born infant after 28 February 2023, is over 4 weeks postpartum, and breastfed for four weeks or longer
* Diagnosed with HIV prior to or during the pregnancy
* If preferred language is other than English, is willing to participate in interviews with an available translator.

Core Activity 1 Inclusion Criteria: Healthcare Providers and Ancillary Healthcare Professionals

* Is of legal age or circumstance to provide independent informed consent
* Is a healthcare provider who self-identifies as an obstetrician, midwife, nurse, adult or pediatric infectious disease specialist, or advance practice provider who participated in the care of at least five PPWH and/or their infants over the three years prior to entry OR
* Is an ancillary healthcare professional who self-identifies as a social worker, lactation support provider, patient navigator, pharmacist, doula who participated in the care of at least five PPWH and/or their infants over the three years prior to entry

Core Activity 1 Inclusion Criteria: Influential Individuals

* Has been identified by a PPWH enrolled in Core Activity 1 as aware of her HIV status and contributing to her infant feeding decisions
* Is of legal age or circumstance to provide independent informed consent
* If preferred language is other than English, is willing to participate in interviews with an available translator.

Core Activity 2 Inclusion Criteria: Pregnant and Postpartum Women with HIV and their Infant

* Is of legal age or circumstance to provide independent informed consent
* Is pregnant with singleton fetus with a gestational age of ≥ 28 0/7 weeks at entry OR
* Gave birth to a live born, singleton infant up to 7 days prior to entry
* Diagnosed with HIV prior to or during the pregnancy
* Expected to be available for the duration of follow-up

Core Activity 3 Inclusion Criteria: Breastfeeding Postpartum Women with HIV and their Infant

* Is of legal age or circumstance to provide independent informed consent
* Must be up to 7 days postpartum with live-born infant
* Diagnosed with HIV prior to or during the pregnancy
* Breastfed her infant for any duration

Core Activity 3 Inclusion Criteria: Pilot Registry Testers

* Is of legal age or circumstance to provide independent informed consent
* Working at a healthcare facility that provides care for women with HIV who are breastfeeding and/or their infants

Exclusion Criteria: Core Activities 1-3

* Has any condition identified during the screening period that, in the opinion of site investigator, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant and postpartum women with HIV (PPWH); healthcare providers (HCP) and ancillary healthcare professionals (AHP) who care for PPWH and/or their infants; other influential individuals who contribute to infant feeding decisions. Pilot registry testers who will enter data into the pilot registry.
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
CA 1: Factors influencing infant feeding decision | Within 28 days and 2 years of Enrollment
  Qualitative themes from in-depth interviews
CA 1: Infants born to women with HIV who receive any breast milk | Monthly, through study completion, up until 5 years
  Binomial outcome from site level surveys
CA 2: Infant feeding method chosen | At 48 weeks post birth
  Binary outcome
CA 2: Breastfeeding initiation among those who intended to breastfeed | At 48 weeks post birth
  Binary outcome
CA 2: Duration of breastfeeding among PPWH who breastfeed | Through 96 weeks post birth
  Numerical outcome
CA 2: Completion of intended duration of breastfeeding | Through 96 weeks post birth
  Binary outcome
CA 2: Mixed method analysis of infant feeding practices from in-depth interviews and survey data | At 48 weeks post birth
  Descriptive joint display table, with qualitative key themes and quantitative findings
CA 2: Breast milk samples with detectable HIV DNA or RNA | Through 48 weeks post birth; At weaning up to 96 weeks post birth
  Binary outcome
CA 2: Viral load measured in different breast milk compartments | Through 48 weeks post birth; At weaning up to 96 weeks post birth
  Numerical outcome
CA 3: Data completed in registry | Through study completion, an average of 3 years
  Binary outcome; whether specified percentage of data is completed in registry
CA 3: Median score on Feasibility of Intervention Measure, Acceptability of Intervention Measure and Appropriateness of Intervention Measures | Through study completion, an average of 3 years
  Numerical outcome
CA 3: Completion of two visit entries for at least three eligible participants | Through study completion, an average of 3 years
  Binary outcome; whether sites complete entries

SECONDARY OUTCOMES:
CA 1: Approaches to support infant feeding decisions and improve quality of care | Within 28 days and 2 years of Enrollment
  Qualitative themes from in-depth interviews
CA 1: Descriptive results of current practices, burden, benefits and resources | Monthly, through study completion, up to 5 years
  Site surveys, provider surveys, In-depth Interviews
CA 2: Median cost per postpartum woman with HIV and infant pair | Through study completion, up to 5 years
  Numerical outcome, by feeding approach
CA 2: Cost effectiveness ratio presented as cost per quality adjusted life year saved in breastfeeding mother/infant pair | Through study completion, up to 5 years
  Numerical outcome
CA 2: Cost per case of medical condition prevented by breastfeeding | Through study completion, up to 5 years
  Numerical outcome
CA 2: Changes in scores of mental health and quality of life surveys | At 20 Weeks, At 48 Weeks
  Numerical outcome, by infant feeding method
CA 2: Satisfaction with infant feeding decision and decision regret survey scores | At 20 weeks, At 48 weeks
  Numerical outcome, by infant feeding method
CA 2: Infant HIV acquisition | Through study completion, up to 96 weeks post birth
  Binary outcome, by infant feeding method
CA 2: Infant weight-for-age, length-for-age, head circumference-for-age (by z-score for sex) | At 20 weeks, At 48 weeks
  Numerical outcome
CA 2: Score classification of each Ages and Stages developmental area | At 20 weeks, At 48 weeks
  Ordinal outcome
CA 2: Plasma HIV viral load | Through 48 weeks post birth, At weaning up to 96 weeks post birth
  Numerical outcome and categorical outcome
CA 2: Number of copies of HIV DNA or RNA per mL of milk | Through 48 weeks post birth, At weaning up to 96 weeks post birth
  Numerical outcome

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Abuogi, Study Chair — University of Colorado, Denver
Locations (11):
- United States (11):
  - University of Southern California (CRS 5048), Los Angeles, California
  - David Geffen School of Medicine at UCLA (CRS 5112), Los Angeles, California
  - University California, San Diego (CRS 4601), San Diego, California
  - University of Colorado, Denver (CRS 5052), Aurora, Colorado
  - University of Florida (5051), Jacksonville, Florida
  - Univ of Miami Pediatric/Perinatal HIV/AIDS (5127), Miami, Florida
  - 5030, Emory University School of Medicine Clinical Research Site, Atlanta, Georgia
  - Lurie Children's Hospital of Chicago (CRS 4001), Chicago, Illinois
  - Johns Hopkins University (CRS 5092), Baltimore, Maryland
  - Jacobi Med. Ctr. Bronx NICHD CRS (5013), The Bronx, New York
  - St. Jude Childrens Research Hosp, Memphis (6501), Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT)
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network and CDC.
  * For what types of analyses? To achieve aims in the proposal approved by the IMPAACT Network and CDC.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https://www.impaactnetwork.org/studies/submit-research-proposal. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data.